CLINICAL TRIAL: NCT04967950
Title: An Efficacy Study of Secukinumab in Enthesitis of Psoriatic Arthritis Patients as Measured by Imaging Test
Brief Title: An Efficacy Study of Secukinumab In Enthesitis of Psoriatic Arthritis Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-IL17
Record Dates: First submitted 2021-07-08; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab; Methotrexate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Secukinumab 300mg (Experimental): Randomized in a 1:1:1 ratio to secukinumab 300mg or secukinumab 150mg or MTX 15mg qw
  Interventions: Drug: Secukinumab 300 MG
- Secukinumab 150mg (Experimental): Randomized in a 1:1:1 ratio to secukinumab 300mg or secukinumab 150mg or MTX 15mg qw
  Interventions: Drug: Secukinumab 150 MG
- methotrexate (Active Comparator): methotrexate
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Secukinumab 300 MG — Secukinumab 150 mg s.c. with loading dose at baseline, week 1,2,3,4 and then every 4 weeks from week 5 up to 12 weeks. After which, if MASEI ultrasound enthesitis score improvement is less than 50%, Secukinumab 150 mg will be with a switch to 300 mg.
  Arms: Secukinumab 300mg
Drug: Secukinumab 150 MG — Methotrexate 15 mg po. every week up to 12 weeks. After which, if MASEI ultrasound enthesitis score improvement is less than 50%, methotrexate with a switch to Secukinumab 150 mg at 12 weeks.
  Arms: Secukinumab 150mg
Drug: Methotrexate — methotrexate
  Arms: methotrexate

SUMMARY:
Given the role of IL-17 in the development of entheseal-driven pathology, a therapeutic strategy aimed at blocking IL-17 would be a logical option for the treatment of enthesitis in psoriatic arthritis patients. This study will be the first randomized trial of a biologic therapy in participants with psoriatic arthritis, using imaging test.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older,;
* had received a diagnosis of psoriatic arthritis at least 6 months previously, fulfilled the Classification Criteria for Psoriatic Arthritis (CASPAR);
* had at least 1 active enthesitis (confirmed by ultrasound) ;
* had active arthritis (at least 3 tender/painful and 3 swollen joints) ;
* had active plaque psoriasis (there was no criteria for minimum psoriasis severity) at screening and baseline.

Exclusion Criteria:

* History of surgery or trauma at the site examined by ultrasound (hand, elbow, knee, ankle, etc.);
* Local injection of glucocorticoids or other drugs at the site examined by ultrasound in recent 6 weeks;
* Peripheral neuropathy;
* Use of IL-17 or IL-12/23 inhibitors in the last 12 months;Use of infliximab, adamumab, golimumab, and cetuzumab in the last 10 weeks;PUVA treatment for the last 4 weeks;Use of topical treatment or UVB phototherapy that may have an effect on psoriasis in the last 2 weeks;
* recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiovascular, or neurologic disease; evidence of active or latent or inadequately treated Mycobacterium tuberculosis; aspartate transaminase (AST) or alanine transaminase (ALT) >3x upper limit of normal (ULN) at screening; estimated creatinine clearance <40 mL/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Madrid Sonographic Enthesis Index (MASEI) ultrasound enthesitis score | Baseline，Week 12 and Week 24
  Twelve entheses will be scored in terms of inflammatory and morphological components according to the OMERACT enthesitis composite semi-quantitative scale (0 to 3). The lowest OMERACT score a participant can have at baseline is 1 (based on Inclusion Criterion, which requires at least 1 points in the B-mode or the Doppler mode in at least one active enthesis ). The highest OMERACT score expected at baseline will be 136, assuming that each of the 12 entheses assessed shows a maximum of 3 points in the gray scale score, and a maximum of 3 points in the Doppler score.

SECONDARY OUTCOMES:
Change from Baseline in the OMERACT Heel Enthesitis MRI Scoring System(HEMRIS) | Baseline and Week 24
  Heel Entheses will be scored in terms of inflammatory and morphological components according to the RAMRIS and PsAMRIS composite semi-quantitative scale (0 to 3). The lowest HEMRIS score a participant can have at baseline is 0. The highest HEMRIS score expected at baseline will be 6, assuming that the heel entheses assessed shows a maximum of 3 points in inflammatory score, and a maximum of 3 points in structure damage.
Change from Baseline in the PsASon13 unilateral ultrasound composite score of synovitis | Baseline，Week 12 and Week 24
  Joints examined by the PsASon13 unilateral ultrasound composite score: Small finger joints: MCP2, MCP5, H-PIP1, H-PIP2, H-PIP3; Distal interphalangeal finger joints: H-DIP3; Small joints of feet: MTP1, MTP5, F-PIP1; Distal interphalangeal joints of feet: F-DIP2, F-DIP3; Large joints: wrist and knee. Lowest score a participant may have at baseline is 0. Highest score a participant may have at baseline is 184 (5 small finger joints, each ranging from 0 to 18; 1 distal interphalangeal finger joint, each ranging from 0 to 16; 3 small joints of feet, each ranging from 0 to 12; 2 distal interphalangeal joints of feet, each ranging from 0 to 12; 1 wrist ranging from 0 to 12; and 1 knee ranging from 0 to 6). Largest change expected from baseline to Week 16 is -118 points (improvement).
Proportion of patients achieving ACR20、ACR50 and ACR70 response. | Baseline，Week 12 and Week 24
  The ACR is a standard criteria originally developed to measure the effectiveness of various arthritis medications or treatments in clinical trials for RA, but is also widely used in PsA. The ACR measures improvement in tender joint count (TJC) or swollen joint count (SJC), and improvement in at least 3 of the following 5 parameters: Patient Global Assessment (PtGA), Physician's Global Assessment of Disease Activity (PhGA), physical function (using HAQ-DI) and acute phase reactant (using CRP). ACR 20 response is achieved if ≥ 20%≥ 50%/≥ 70% improvement in tender joint count (TJC) or swollen joint count (SJC) as well as a ≥ 20%/≥ 50%/≥ 70% improvement in ≥ 3 of the other 5 parameters.
Number of participants who achieve Psoriasis Area and Severity Index 75 (PASI 75) | Baseline，Week 12 and Week 24
  Scores range from 0 to 72. A score of more than 10 generally translates to "moderate-to-severe". Usually, the higher your PASI score, the lower the quality of life. A PASI 75 is at least a 90% improvement (reduction) in PASI score.
Change from Baseline in Dermatology Life Quality Index (DLQI) score | Baseline and Week 24
  A 10-item measure to assess health-related quality of life in adults with skin diseases. Scores range from 0-30 with a higher score being less quality of life.
Change from Baseline in HAQ-DI score | Baseline and Week 24
  Health Assessment Questionnaire-Disability Index (HAQ-DI) is a 20-question scale assessing functional ability. The final HAQ-DI score ranges from 0 (no problems functioning) to 3 (not able to function).

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided